CLINICAL TRIAL: NCT01082627
Title: Prospective, Multi-centers, Investigator Sponsored, Randomized Controlled Trial Towards Identifying the Effect of Somatostatin Treatment in Early Postoperative Simple Small Bowel Obstruction
Brief Title: Identifying the Effect of Somatostatin Treatment in Early Postoperative Simple Small Bowel Obstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nanjing PLA General Hospital (Other)
Responsible Party: NLi, Nanjing Jinling Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Nanjing Jinling Hospital
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2010-02

CONDITIONS: Small Bowel Obstruction
Keywords: Somatostatin small bowel obstruction
MeSH Terms: interventions — Somatostatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Somatostatin+common daily practice (Experimental)
  Interventions: Drug: Somatostatin
- common daily practice (Placebo Comparator)
  Interventions: Other: common daily practice

INTERVENTIONS:
Drug: Somatostatin — 250ug/h,Continuous I.V. infusion,maximal 14 days
  Other Names: Stilamin
  Arms: Somatostatin+common daily practice
Other: common daily practice — common daily practice
  Arms: common daily practice

SUMMARY:
Primary Objective:

To demonstrate whether an early fixed Somatostatin treatment improves the complete recovery rate of early postoperative simple small bowel obstruction (EPSSBO) compared with the common daily practice

Notes:

1. complete recovery= toleration of solid food+ flatus+ passage+ recovery of bowel movement.
2. common daily practice includes:

   * NPO (Nil per mouth), re-dehydration, TPN (Total Parenteral Nutrition) if needed. Check & make sure stability of electrolytes daily.
   * GI (Gastro-Intestinal) depression via NGT (Naso-Gastric Tube)
   * Discontinue opiates, instead of NSAIDs. (Non-Steroidal Anti-Inflammatory Drugs)
   * Pro-dynamic drugs or other drugs which may interfere with GI (Gastro-Intestinal) movement eg. anti-histamines, anti-cholinergic, opiates, anti-depressives are not indicated.

Secondary Objectives:

To investigate whether an early fixed Somatostatin treatment will bring much benefit to EPSSBO pts compared with the common daily practice,for this purpose,the study will investigate the endpoints below.

DETAILED DESCRIPTION:
1. Study Design:

   This is a multi-centers, open label, randomized study , and will enroll 80 EPSSBO patients, who will be assigned to two groups randomly. All the inclusive patients will be consistent with the diagnosis of EPSSBO, and the mechanic SBO or the strangulating SBO will be ruled out in advance.

   The inclusive patients will be assigned to two groups as follow(ratio 3:1)
   * Arm A: Somatostatin+common daily practice(60).
   * Arm B: common daily practice only(20).
2. Total number of subjects:80 EPSSBO patients.
3. Schedule of visits and assessments,The following assessments will be performed.

   * Pre-screening:informed consent,demographic data,EPSSBO diagnosis.
   * Screening
   * Daily visit:
   * Weekly visit：
   * End of study visit：
4. Statistical methods

   * As this will be a pilot study, no formal statistical calculations were carried out and the sample size was estimated as 80 EPSSBO subjects in a 3:1 ratio of active to control subjects i.e. 60 for Stilamin+ common daily practice and 20 for common daily practice only.
   * The primary endpoint of the complete recovery rate will be estimated for both treatment groups, with 95% confidence intervals. The difference in the proportions between the treatment groups will also be estimated and treatment comparisons will be performed using a chi-square test. All statistical tests will be 2-tailed with a significance level of 0.05.
   * Descriptive statistics including number (N), mean, median, standard deviation, minimum and maximum, will be produced for all continuous variables. Frequency tables of number (N) and percentage of subjects will be produced for all categorical variables.
   * Continuous variables will be analyzed using an analysis of variance (ANOVA) model with effect for treatment only. The data will be checked for normality. If the distributions are normal, parametric techniques will be used. If the data are not normally distributed, non parametric techniques will be used. These assumptions will also apply to the primary endpoint i.e. use of non-parametric tests if necessary. All statistical tests will be 2-tailed with a significance level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Patient has given written informed consent before any study-related activities are carried out.
* Males and females,aged 18-70.
* Recent open abdominal surgery history.
* Having the following symptoms or signs after 5 days of index operation: abdominal distention + inability to pass flatus + inability to passage + weak or absent bowel sound.
* X-ray:paucity of bowel gas,0-1 air-fluid level.
* CT:intestinal wall edema/thickness,no mechanic obstruction

Exclusion Criteria:

* After laparoscopic surgery.
* Recent drug history of anti-histamines,anti-cholinergic,anti-depressives,post-operative usage of opiates.
* Any of below:severe abdominal pain,colic,peritoneal sign,hig-pitched bowel sound,T>38℃,tachycardia,bradycardia,WBC>12000/ul,X-ray≥2 air-fluid levels,CT:mechanic obstruction.
* Any of below: Abdominopelvic abscess,Anastomotic leaks, Appendicitis,Cholecystitis,Hemoperitoneum or retroperitoneal hemorrhage, Hypokalemia, Hypomagnesemia, Pancreatitis, Sepsis.Uremia.
* Severe heart failure（NYHA III and above）.
* History of arrhythmia or syncope.
* ECG QTc >0.44s.
* Severe renal function insufficiency （Calculated Creatinine Clearance Rate (Ccr) <30ml/min）.
* Severe Liver function insufficiency（CHILD B~C）.
* Hyper or hypothyroidism intracranial GH-secreting tumor.
* Brittle DM.
* Pregnancy.
* Allergy to any ingredient of Stilamin.
* History of significant neurologic or psychiatric disorders including dementia, seizures, bipolar disorder.
* Medical or psychological condition that would not permit the patient to complete the study or sign the informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2009-06; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Complete recovery rate of EPSSBO = (Num. of patients with complete recovery of EPSSBO per group/Total num. of patients per group) * 100 | 14 days

SECONDARY OUTCOMES:
Average recovery time | 14 days
Re-surgery rate | 14 days
Average NG (naso-gastric) aspirate volume | 14 days
Average re-dehydration volume | 14 days
Change of blood electrolytes | 14 days
Degree of symptom and sign relief | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing PLAGH, Nanjing, Jiangsu, China